CLINICAL TRIAL: NCT05931068
Title: Pre- and Postoperative Energy Expenditure in Major Liver Resection: What do we Ask From a Patient?
Brief Title: Perioperative Energy Expenditure in Major Liver Resection
Acronym: PRO-NRG
Status: Recruiting | Type: Observational
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, Nicole Hildebrand, Coordinating Investigator, Academisch Ziekenhuis Maastricht
Other Study IDs: NL78760.068.21
Record Dates: First submitted 2023-05-04; First posted 2023-07-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Liver Diseases; Liver Neoplasms
Keywords: Energy expenditure; Aerobic capacity; Resting metabolism rate; Metabolic demand; Physical activity; Pre- and post-operative assessment
MeSH Terms: conditions — Neoplasms; Liver Diseases; Liver Neoplasms; Motor Activity | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pre- and postoperative assessment — Pre- and postoperative assessment will consist of measurement of energy expenditure (direct and indirect calorimetry), aerobic capacity (cardiopulmonary exercise test), and physical activity (accelerometry).

SUMMARY:
Rationale: Complication rates after major liver resections remain as high as 43%. Many initiatives have been taken to reduce postoperative morbidity. As such, prehabilitation programmes are increasingly used for patients undergoing major abdominal surgery. Improvement of aerobic fitness has been proven to reduce complication rates, especially in high-risk patients (those with a low preoperative aerobic capacity). Different conceptual hypotheses exist of the underlying mechanism of variability in postoperative complications and prehabilitation response. One of the complementary rationales focusses on homeostasis-allostasis before and after surgery, more specifically on the preoperative aerobic capacity to meet postoperative metabolic demands. However, more insight in postoperative metabolic demands (energy expenditure) during in-hospital recovery from major abdominal surgery in relation to preoperative resting metabolic demands and maximal aerobic capacity is essential to understand the increase in metabolic demands coinciding with major surgery in relation to the body's reserve capacity. This information can be used to better understand the rationale behind exercise prehabilitation, as well as to optimize the content of preoperative treatment for unfit patients, for instance by means of personalized prehabilitation programs that might improve postoperative outcomes.

Objective: This study aims to explore the difference of pre- and postoperative energy expenditure in patients undergoing major elective liver resection and relate this to their preoperative aerobic capacity.

Study design: The study will be a prospective observational study with thorough pre- and postoperative measurements of energy expenditure. Energy expenditure will be measured using the doubly labelled water method, as well as by indirect calorimetry. To assess aerobic capacity, cardiopulmonary exercise testing will be performed pre- and postoperatively. Additionally, accelerometers will be used to evaluate pre- and postoperative physical activity levels.

Study population: Patients aged ≥18 years undergoing major liver resection (≥3 segments) will be asked to participate. The inability to perform cardiopulmonary exercise testing, neo-adjuvant chemotherapy, and cirrhotic liver are reasons for exclusion.

Main study parameters/endpoints: The main study parameter is the difference of energy expenditure pre- and postoperatively, as measured with doubly labelled water and indirect calorimetry.

Secondary endpoints: Additionally, as secondary endpoints, aerobic fitness, physical activity level, and postoperative complications will be assessed.

DETAILED DESCRIPTION:
The number of major surgical procedures performed in older patients has been rising in recent years. Older-aged patients have a higher risk of postoperative morbidity and mortality. A recent Dutch study reported that 43% of the patients had a complicated postoperative course after major liver resection (≥3 segments) performed for colorectal liver metastases. The risk of postoperative complications and mortality is related to the patient's age combined with a higher prevalence of comorbidities, which both decrease the physiological reserve capacity of organ systems. As such, preoperative aerobic capacity has been found to be independently and consistently associated with postoperative outcomes after liver surgery. Interestingly, exercise prehabilitation is known to preoperatively increase the aerobic fitness of patients scheduled for major elective abdominal surgery. High-risk patients will benefit most from this, with a reduction in postoperative complications of >30%.

The conceptual hypothesis of exercise prehabilitation as part of perioperative care in patients undergoing major abdominal surgery is clear and increasingly substantiated with evidence. However, when taking into account the variation in prehabilitation programs and the variability of individual prehabilitation outcomes, there is room for improvement by exploring different rationales subserving the conceptual hypothesis of prehabilitation. One of the complementary rationales focusses on homeostasis-allostasis before and after surgery, more specifically on the preoperative metabolic capacity to meet postoperative metabolic demands. However, more insight in postoperative metabolic demands (energy expenditure) during in-hospital recovery from major abdominal surgery in relation to preoperative resting metabolic demands and maximal aerobic capacity is essential to understand the increase in metabolic demands coinciding with major surgery in relation to the body's reserve capacity. Insight in this can subsequently be used to further optimize the content of preoperative preventive interventions for unfit patients (exercise prehabilitation) to improve patient- and treatment-related outcomes.

Study design:

This study will be an explorative prospective observational cohort study of 18 months, in which energy expenditure will be determined pre- and postoperatively in 20 patients undergoing major elective liver resection at the Maastricht University Medical Center+ (MUMC+). Patients undergoing major liver resection (≥3 segments) were chosen for this study given the magnitude of their surgery and high prevalence of postoperative morbidity.

This is a monocenter study, where all measurements will be performed at the Clinical Research Unit of the MUMC+. Energy expenditure will be quantified one week before and one week after surgery using the doubly labelled water (DLW) technique, as well as by using indirect calorimetry measurements during the hospital admission one day before surgery, at postoperative day 1, 2, and 3, and at hospital discharge. Moreover, aerobic capacity will be determined with cardiopulmonary exercise testing (CPET) preoperatively and at hospital discharge.

Study procedures:

Doubly labelled water Energy expenditure over the week prior to surgery and the week after surgery will be measured using the doubly labelled water (DLW) technique. Subjects receive a dose of DLW at one time point, that is, one week before surgery. The given dose (2.5 g/L total body water (TBW) of a water mixture containing 9.8% enriched H218O and 6.5% enriched 2H2O) will be calculated based on the subject's TBW, which will be estimated based on age, sex, and BMI. Baseline urine samples will be collected prior to dosing (-8 days). After overnight equilibration, the second urine sample will be collected from the second morning urine. Subsequent urine samples will be collected the evening before surgery, just prior to incision in the operating room, at discharge, and if feasible at the end of the observation period, which will cover one week preoperatively and one week postoperatively or up until hospital discharge if admission is shorter than 7 days. Urine samples will be collected and stored at -20C at the hospital. All urine samples will be transported to Maastricht University for storage until analysis to evaluate energy expenditure, for which the Maastricht protocol will be used.

Indirect calorimetry Resting energy expenditure on the day before surgery (hospital admission), at postoperative day 1, 2, and 3, and at hospital discharge will be determined using indirect calorimetry. A subject's resting metabolic rate (RMR) will be determined in the morning after an overnight fast in a thermoneutral environment. Using a ventilated hood system (Q -NRG, COSMED, Rome, Italy), RMR will be measured for 10 minutes while the subject is lying in their bed. To eliminate habituation effects and reach complete resting conditions, respiratory measurements collected during the first 5 minutes will be discarded, and the remaining 5 minutes will be used to calculate RMR. The machine analyses inspired and expired air samples within a micro-mixing chamber. Mean values of VO2, VCO2, and energy expenditure (EE) are given. Every month, the ventilated hood system will be calibrated according to factory guidelines.

Aerobic capacity To assess a subject's aerobic capacity, CPET up to volitional exertion will be performed on a cycle ergometer (Lode Corival, Lode BV, Groningen) one week before hospital admission and at hospital discharge. Expectedly, the majority of patients will be able to undergo maximal CPET at discharge. At the time of discharge any major complication that occurred during hospital admission, will have been resolved. If the patient does not feel fit for maximal CPET, patients will have the ability to choose to either perform submaximal CPET, or no CPET at hospital discharge. During CPET, subjects breathe through a facemask connected to a calibrated ergo spirometry system (Vyntus CPX, Vyaire Medical, Hoechberg). Breath-by-breath minute ventilation, VO2, and VCO2 will be calculated and averaged at 10-second intervals. Heart rate will be measured by continuous 12-lead electrocardiography. Peak VO2 (VO2peak) will be calculated as the average value over the last 30 seconds before termination of the test. The VO2 at the ventilatory anaerobic threshold will be determined using the modified V-slope method. The preoperative and postoperative CPET will be performed in presence of an experienced investigator and physician.

Maximal CPETs will be performed using a calibrated electronically braked cycle ergometer pre- and post-intervention at the hospital. The patient will be fitted with a 12-lead electrocardiogram to measure heart rate and heart rhythm, as well as with a face mask (7450 V2, Hans Rudolph Inc, Kansas City, MO, USA) connected to a calibrated respiratory gas analysis system that will calculate breath-by-breath VO2, carbon dioxide production, and minute ventilation throughout the CPET. Gas analyzers will be calibrated using gases of known concentration, whereas the flow meter will be calibrated using a three-liter syringe. Blood pressure will be monitored, and peripherally measured oxygen saturation will be measured at the index finger. Each patient will be carefully instructed, where after he or she will be fitted with all equipment.

After two minutes of rest measurements, the patient starts cycling at a workload of 0 W (unloaded). Patients will be instructed to maintain a pedaling frequency of around 80 revolutions per minute throughout the test. After three minutes of unloaded cycling, work rate will be linearly incremented with a 5, 10, 15, or 20 W/min ramp protocol (depending on the patient's physical fitness to ensure a test duration between eight and twelve minutes) until the patient stops due to volitional exhaustion, despite strong verbal encouragement. Test effort will be considered maximal when the participant shows objective (a heart rate at peak exercise >95% of predicted and/or a respiratory exchange ratio at peak exercise >1.10) and subjective (unsteady biking, sweating, facial flushing, and clear unwillingness to continue despite encouragement) signs of a maximal effort. Peak exercise is defined as the point at which the pedaling frequency falls definitely <60 revolutions per minute. Heart rate, VO2, carbon dioxide production, work rate, minute ventilation, peripherally measured oxygen saturation, and pedaling frequency will be measured continuously during the baseline measurements, unloaded cycling, ramp-protocol, and a three-minute recovery phase at 25 W. Output from the metabolic test system, including heart rate, VO2, carbon dioxide production, minute ventilation, and pedaling frequency will be averaged at ten-second intervals and stored for further use. In order to measure the level of perceived exertion before and directly after CPET, a 6-20 Borg scale for rating of perceived exertion will be used. The perception of exertion is mainly felt as strain and fatigue in the patient's muscles and breathlessness.

CPET parameters will be averaged into 10-second intervals after outliers (>3 standard deviations from the local mean) are removed. CPET interpretation will be performed by a trained and experienced clinical exercise physiologist. Absolute values at peak exercise (e.g., VO2peak) will be calculated as the average value over the last 30 seconds before termination of the test. Peak heart rate is defined as the highest heart rate achieved during the test. The ventilatory anaerobic threshold is defined as the point at which the ventilatory equivalent for oxygen and the partial end-tidal oxygen tension reached a minimum and thereafter began to rise in a consistent manner, coinciding with an unchanged ventilatory equivalent for carbon dioxide and partial end-tidal carbon dioxide tension. When this ventilatory equivalents method appeared to provide uncertain results for a patient's ventilatory anaerobic threshold, the point at which the linear slope of the relation between the carbon dioxide production and oxygen uptake changed was taken as the ventilatory anaerobic threshold, according to the V-slope method. The ventilatory anaerobic threshold will be expressed as an absolute and relative value (normalized for body mass). The graphical presentation of the minute ventilation as a function of carbon dioxide production during the incremental cardiopulmonary exercise test will be used to determine the point at which the minute ventilation increased out of proportion to carbon dioxide production, that is, the respiratory compensation point. The slope of the relationship between the minute ventilation and carbon dioxide production will be calculated by linear least squares regression of the relation between the minute ventilation and carbon dioxide production up to the respiratory compensation point.

Accelerometry Accelerometers will be used to monitor body movement, representing physical activity. From that variability in physical activity between days can be monitored. The accelerometer used is the MOX accelerometer (Maastricht Instruments, Maastricht, The Netherlands), which measures only 35 x 35 x 10 mm and weighs 11 gr. Because of this small size and weight, this accelerometer does not to interfere with daily activities and does not pose a burden to subjects. The sensor will be attached via a plaster on the upper thigh, 10 centimeters above the knee. The adhesive plaster will be attached in the presence of an investigator. At the time of hospital admission, and after surgery, the position of the adhesive plaster will be checked and adjusted if necessary. Patients will receive their accelerometer after aerobic fitness testing and hand it in right before the last aerobic fitness testing. The device contains a tri-axial accelerometer sensor that stores the data within the device. Data will be analyzed offline, and can be classified as sedentary, standing, or physical active. It has been validated in hospitalized patients, elderly, and cancer survivors.

Hospital anxiety and depression scale questionnaire Depressive symptoms might be associated with decreased physical activity and energy expenditure. Given that depressive symptoms are common in cancer patients, it could be a possible confounder when estimating daily physical activity. Therefore, subjects will be screened using the hospital anxiety and depression scale (HADS). This is a well-validated scale specifically for non-psychiatric patients with physical illness. The scale has been validated for chronically ill patients as well as oncology patients and consists of 14 questions on depressive (7 questions) and anxiety symptoms (7 questions) with a range of 0 to 3. A score of 8 or higher in either subset indicates a possible anxiety of depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Scheduled for open liver resection (≥3 segments) at the MUMC+
* Able to understand the Dutch language sufficiently to give consent and follow orders during study assessments

Exclusion Criteria:

* Cirrhotic liver
* Unable or unwilling to perform CPET or indirect calorimetry
* Liver ablation as the primary treatment
* Termination of surgery due to too extensive oncological disease (open-close surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults, requiring major liver resection (≥3 segments) for any kind of malignant indication at Maastricht UMC+
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in energy expenditure using direct calorimetry | through monitoring period, average of 2 weeks perioperatively
  Direct calorimetry applying the doubly labelled water method
Change in energy expenditure using indirect calorimetry | through monitoring period, average of 2 weeks perioperatively
  Indirect calorimetry applying a ventilated hood system

SECONDARY OUTCOMES:
Preoperative aerobic fitness | One week prior to surgery
  Estimation of aerobic fitness using the gold standard of cardiopulmonary exercise testing, expressed as the maximal oxygen uptake (VO2) at the ventilatory anaerobic threshold
Postoperative aerobic fitness | end of monitoring period, average of 2 weeks postoperatively
  Estimation of aerobic fitness using the gold standard of cardiopulmonary exercise testing, expressed as the maximal oxygen uptake (VO2) at the ventilatory anaerobic threshold
Perioperative physical activity level | through monitoring period, average of 2 weeks perioperatively
  Accelerometry data of tri-axial movement
Postoperative complications | 30-day postoperatively
  Postoperative complications rated according to Clavien-Dindo classification
Liver-specific postoperative complications | 30-day postoperatively
  bile leakage, post-resection liver failure or intra-abdominal abscess
Length of hospital stay | Through study completion, an average of 10 days
  Time between surgery and postoperative hospital discharge in days
Hospital anxiety and depression scale | Baseline (At the beginning of monitoring period)
  Using the "Hospital anxiety and depression scale"-questionnaire, consisting of 14 questions on depressive (7 questions) and anxiety (7 questions) symptoms

CONTACTS AND LOCATIONS:
Overall Officials: S.W.M. Olde Damink, MD MSc PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lu Q, Lu JW, Wu Z, Liu XM, Li JH, Dong J, Yin GZ, Lv Y, Zhang XF. Perioperative outcome of elderly versus younger patients undergoing major hepatic or pancreatic surgery. Clin Interv Aging. 2018 Jan 24;13:133-141. doi: 10.2147/CIA.S153058. eCollection 2018. PMID 29416321
- [Background] van der Werf LR, Kok NFM, Buis CI, Grunhagen DJ, Hoogwater FJH, Swijnenburg RJ, den Dulk M, Dejong KCHC, Klaase JM; Dutch Hepato Biliary Audit Group. Implementation and first results of a mandatory, nationwide audit on liver surgery. HPB (Oxford). 2019 Oct;21(10):1400-1410. doi: 10.1016/j.hpb.2019.02.021. Epub 2019 Mar 26. PMID 30926330
- [Background] Wilson RJ, Davies S, Yates D, Redman J, Stone M. Impaired functional capacity is associated with all-cause mortality after major elective intra-abdominal surgery. Br J Anaesth. 2010 Sep;105(3):297-303. doi: 10.1093/bja/aeq128. Epub 2010 Jun 23. PMID 20573634
- [Background] Moran J, Wilson F, Guinan E, McCormick P, Hussey J, Moriarty J. Role of cardiopulmonary exercise testing as a risk-assessment method in patients undergoing intra-abdominal surgery: a systematic review. Br J Anaesth. 2016 Feb;116(2):177-91. doi: 10.1093/bja/aev454. PMID 26787788
- [Background] Junejo MA, Mason JM, Sheen AJ, Moore J, Foster P, Atkinson D, Parker MJ, Siriwardena AK. Cardiopulmonary exercise testing for preoperative risk assessment before hepatic resection. Br J Surg. 2012 Aug;99(8):1097-104. doi: 10.1002/bjs.8773. Epub 2012 Jun 14. PMID 22696424
- [Background] Thomas G, Tahir MR, Bongers BC, Kallen VL, Slooter GD, van Meeteren NL. Prehabilitation before major intra-abdominal cancer surgery: A systematic review of randomised controlled trials. Eur J Anaesthesiol. 2019 Dec;36(12):933-945. doi: 10.1097/EJA.0000000000001030. PMID 31188152
- [Background] Dunne DF, Jack S, Jones RP, Jones L, Lythgoe DT, Malik HZ, Poston GJ, Palmer DH, Fenwick SW. Randomized clinical trial of prehabilitation before planned liver resection. Br J Surg. 2016 Apr;103(5):504-12. doi: 10.1002/bjs.10096. Epub 2016 Feb 11. PMID 26864728
- [Background] Bongers BC, Punt IM, van Meeteren NL. On "Prehabilitation: The emperor's new clothes or a new arena for physical therapists?" Lundberg M, Archer KR, Larsson C, Rydwik E. Phys Ther. 2018;12:127-130. Phys Ther. 2019 Jul 1;99(7):953-954. doi: 10.1093/ptj/pzz064. No abstract available. PMID 31108508
- [Background] West MA, Wischmeyer PE, Grocott MPW. Prehabilitation and Nutritional Support to Improve Perioperative Outcomes. Curr Anesthesiol Rep. 2017;7(4):340-349. doi: 10.1007/s40140-017-0245-2. Epub 2017 Nov 7. PMID 29200973
- [Background] Goldstein DS, McEwen B. Allostasis, homeostats, and the nature of stress. Stress. 2002 Feb;5(1):55-8. doi: 10.1080/102538902900012345. PMID 12171767
- [Background] Bongers BC, Dejong CHC, den Dulk M. Enhanced recovery after surgery programmes in older patients undergoing hepatopancreatobiliary surgery: what benefits might prehabilitation have? Eur J Surg Oncol. 2021 Mar;47(3 Pt A):551-559. doi: 10.1016/j.ejso.2020.03.211. Epub 2020 Mar 29. PMID 32253075
- [Background] Deurenberg P, Weststrate JA, Seidell JC. Body mass index as a measure of body fatness: age- and sex-specific prediction formulas. Br J Nutr. 1991 Mar;65(2):105-14. doi: 10.1079/bjn19910073. PMID 2043597
- [Background] Westerterp KR, Wouters L, van Marken Lichtenbelt WD. The Maastricht protocol for the measurement of body composition and energy expenditure with labeled water. Obes Res. 1995 Mar;3 Suppl 1:49-57. doi: 10.1002/j.1550-8528.1995.tb00007.x. PMID 7736290
- [Background] Delsoglio M, Dupertuis YM, Oshima T, van der Plas M, Pichard C. Evaluation of the accuracy and precision of a new generation indirect calorimeter in canopy dilution mode. Clin Nutr. 2020 Jun;39(6):1927-1934. doi: 10.1016/j.clnu.2019.08.017. Epub 2019 Sep 10. PMID 31543335
- [Background] Levett DZH, Jack S, Swart M, Carlisle J, Wilson J, Snowden C, Riley M, Danjoux G, Ward SA, Older P, Grocott MPW; Perioperative Exercise Testing and Training Society (POETTS). Perioperative cardiopulmonary exercise testing (CPET): consensus clinical guidelines on indications, organization, conduct, and physiological interpretation. Br J Anaesth. 2018 Mar;120(3):484-500. doi: 10.1016/j.bja.2017.10.020. Epub 2017 Nov 24. PMID 29452805
- [Background] Lamarra N, Whipp BJ, Ward SA, Wasserman K. Effect of interbreath fluctuations on characterizing exercise gas exchange kinetics. J Appl Physiol (1985). 1987 May;62(5):2003-12. doi: 10.1152/jappl.1987.62.5.2003. PMID 3110126
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Beaver WL, Wasserman K, Whipp BJ. A new method for detecting anaerobic threshold by gas exchange. J Appl Physiol (1985). 1986 Jun;60(6):2020-7. doi: 10.1152/jappl.1986.60.6.2020. PMID 3087938
- [Background] Bijnens W, Aarts J, Stevens A, Ummels D, Meijer K. Optimization and Validation of an Adjustable Activity Classification Algorithm for Assessment of Physical Behavior in Elderly. Sensors (Basel). 2019 Dec 4;19(24):5344. doi: 10.3390/s19245344. PMID 31817164
- [Background] van Dijk-Huisman HC, Bijnens W, Senden R, Essers JMN, Meijer K, Aarts J, Lenssen AF. Optimization and Validation of a Classification Algorithm for Assessment of Physical Activity in Hospitalized Patients. Sensors (Basel). 2021 Feb 27;21(5):1652. doi: 10.3390/s21051652. PMID 33673447
- [Background] van Roekel EH, Winkler EA, Bours MJ, Lynch BM, Willems PJ, Meijer K, Kant I, Beets GL, Sanduleanu S, Healy GN, Weijenberg MP. Associations of sedentary time and patterns of sedentary time accumulation with health-related quality of life in colorectal cancer survivors. Prev Med Rep. 2016 Jul 1;4:262-9. doi: 10.1016/j.pmedr.2016.06.022. eCollection 2016 Dec. PMID 27419042
- [Background] Wielopolski J, Reich K, Clepce M, Fischer M, Sperling W, Kornhuber J, Thuerauf N. Physical activity and energy expenditure during depressive episodes of major depression. J Affect Disord. 2015 Mar 15;174:310-6. doi: 10.1016/j.jad.2014.11.060. Epub 2014 Dec 8. PMID 25532078
- [Background] Mitchell AJ, Chan M, Bhatti H, Halton M, Grassi L, Johansen C, Meader N. Prevalence of depression, anxiety, and adjustment disorder in oncological, haematological, and palliative-care settings: a meta-analysis of 94 interview-based studies. Lancet Oncol. 2011 Feb;12(2):160-74. doi: 10.1016/S1470-2045(11)70002-X. Epub 2011 Jan 19. PMID 21251875
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Annunziata MA, Muzzatti B, Bidoli E, Flaiban C, Bomben F, Piccinin M, Gipponi KM, Mariutti G, Busato S, Mella S. Hospital Anxiety and Depression Scale (HADS) accuracy in cancer patients. Support Care Cancer. 2020 Aug;28(8):3921-3926. doi: 10.1007/s00520-019-05244-8. Epub 2019 Dec 19. PMID 31858249
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252